CLINICAL TRIAL: NCT04483947
Title: A Phase 1, Double Blind, Randomised, Placebo-Controlled, Multi-centre, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD2693 in Patients With Non-alcoholic Steatohepatitis (NASH) With Fibrosis Stage 0-3 and Carriers of the PNPLA3 148M Risk Alleles
Brief Title: A Study to Assess Safety, Tolerability, PK and PD of AZD2693 in Non-alcoholic Steatohepatitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D7830C00002
Record Dates: First submitted 2020-07-06; First posted 2020-07-23 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: Pharmacokinetics; Pharmacodynamics; Obese; PNPLA3 148M Risk Alleles; Multiple Ascending Dose
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be blinded for all study site personal including the principal investigator during the clinical conduct of a given cohort. Investigators will remain blinded to each participant's assigned study intervention throughout the course of the study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort 1 (Experimental): 15 participants will receive AZD2693 dose 1 and 5 participants will receive placebo
  Interventions: Drug: AZD2693; Other: Placebo
- Cohort 2 (Experimental): 15 participants will receive AZD2693 dose 2 and 5 participants will receive placebo
  Interventions: Drug: AZD2693; Other: Placebo
- Cohort 3 (Experimental): 15 participants will receive AZD2693 dose 1 and 5 participants will receive placebo
  Interventions: Drug: AZD2693; Other: Placebo
- Cohort 4 (Experimental): 15 participants will receive AZD2693 dose 3 and 5 participants will receive placebo
  Interventions: Drug: AZD2693; Other: Placebo

INTERVENTIONS:
Drug: AZD2693 — Subcutaneous administration of AZD2693 multiple ascending doses in participants with NASH and who are carriers of the PNPLA3 148M risk allele(s).
Other: Placebo — Participants randomised to placebo will receive the corresponding dose volume of solution as participants receiving AZD2693 within the same cohort

SUMMARY:
This study is intended to investigate the safety and tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of AZD2693, following subcutaneous (SC) administration of multiple ascending doses in participants with Non-alcoholic Steatohepatitis (NASH) with fibrosis Stage 0 to 3 and who are carriers of the patatin-like phospholipase domain-containing 3 (PNPLA3) 148M risk alleles.

DETAILED DESCRIPTION:
This study is a double blind, randomised, placebo-controlled, multi-centre study in participants with NASH and fibrosis stage between F0 (no fibrosis) and F3 (bridging fibrosis), and who are carriers of the PNPLA3 148M risk alleles.

The study will comprise of:

* An optional Pre-Screening Visit may be completed to determine PNPLA3 genotype and collect minimal baseline data and participants who are carriers of the PNPLA3 148M risk allele(s) will continue the study and enter the Screening Period.
* A Screening Period with a maximum of 60 days.
* For participants in all Cohorts, the dosing period will be 8 weeks during which participants will be resident of the study site for Dose 1 and Dose 3. Dose 1 will have participants reside at the study site from the day prior to study intervention administration (Day -1) until at least 2 days after study intervention administration with discharge on Day 3. Dose 2 will be administered at the study site on Day 29 with no overnight stay. Dose 3 will have participants reside at the study site from the day prior to study intervention administration (Day 56) until at least 2 days after study intervention administration with discharge on Day 59.
* Each participant will be followed for approximately 15 weeks post last dose.

The study will be performed at up to 30 study sites in the United States (US) and up to 5 study sites in Mexico. Approximately 80 participants comprising of male and female participants of non-childbearing potential may be enrolled into the first 4 cohorts of this study in order to achieve a target of 56 to 64 evaluable participants.

ELIGIBILITY:
Inclusion Criteria:

For Cohorts 1 to 3:

* An MRI-PDFF ≥7% and one of the following:

  * Previous liver biopsy: Acceptable if taken in the previous 3 years for fibrosis stages F0 to F2, or within the previous 1 year for stage F3; or
  * Previous imaging results taken in the previous 2 years: An MRE between 2.55 kPa and 3.63 kPa, or a vibration-controlled transient elastography (VCTE) between 7.1 kPa and 11.9 kPa;
* Participants who are homozygous for rs738409 (PNPLA3 148M). Cohort 2 will enroll participants who are heterozygous for PNPLA3 148M.

For Cohort 4:

• An MRI-PDFF ≥ 7% and participant's consent for a liver biopsy.

* Participants with suspected or confirmed Non-alcoholic fatty liver disease (NAFLD) or NASH are eligible for the Screening liver biopsy if they meet main protocol inclusion/exclusion criteria AND have any of the following:

Alanine aminotransferase > Upper Limit of Normal (ULN) but < 3 × ULN, OR Imaging demonstrating hepatic steatosis including attenuation parameter (CAP) > 290dB/m, OR A Magnetic resonance elastography (MRE) between 2.55 kPa and 3.63 kPa, or a vibration-controlled transient elastography (VCTE) between 7.1 kPa and 11.9 kPa.

* Histologic evidence of NAFLD or NASH with a NASH Activity Score (NAS) ≥ 3 (independent of subcategory scoring) following Screening liver biopsy.
* Participants who are homozygous for rs738409 (PNPLA3 148M).

Exclusion Criteria:

* History of liver transplant, or current placement on a liver transplant list (this may be checked at the optional Pre-Screening Visit).
* History or presence of hepatic disease (with the exception of hepatic steatosis, NASH) or evidence of other known forms of known chronic liver disease such as alcoholic liver disease, hepatitis B, primary biliary cirrhosis, primary sclerotic cirrhosis, autoimmune hepatitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug-induced liver injury, known or suspected hepatocellular carcinoma (this may be checked at the optional Pre-Screening Visit).
* Histological or imaging (MRE or VCTE) evidence of cirrhosis.
* Participants with history or pre-existing renal disease, as defined below:

  - estimated glomerular filtration rate < 60 mL/min/1.73 m^2 (calculated using the Chronic Kidney Disease Epidemiology Collaboration formula)
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds).
* History of major bleed or high-risk of bleeding diathesis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 32 weeks (From Screening to Final Visit)

SECONDARY OUTCOMES:
Absolute change from baseline to Week 8 and Week 12 in liver fat content (LFC) | Baseline (Day 1), Week 8, Week 12
Percent change from baseline to Week 8 and Week 12 in liver fat content (LFC) | Baseline (Day 1), Week 8, Week 12
Absolute change from baseline in Alanine Aminotransferase | Up to 32 weeks (From Pre-Screening to Final Visit)
Percent change from baseline in Alanine Aminotransferase | Up to 32 weeks (From Pre-Screening to Final Visit)
Absolute change from baseline in Aspartate Aminotransferase | Up to 32 weeks (From Pre-Screening to Final Visit)
Percent change from baseline in Aspartate Aminotransferase | Up to 32 weeks (From Pre-Screening to Final Visit)
Absolute change from baseline in Gamma Glutamyl Transferase | Up to 32 weeks (From Pre-Screening to Final Visit)
Percent change from baseline in Gamma Glutamyl Transferase | Up to 32 weeks (From Pre-Screening to Final Visit)
Absolute change from baseline in Enhanced Liver Fibrosis (ELF) score | Up to 32 weeks (From Pre-Screening to Final Visit)
Percent change from baseline in ELF score | Up to 32 weeks (From Pre-Screening to Final Visit)
Absolute change from baseline in plasma pharmacodynamic biomarker | Days 1, 8, 29, 36, 50, 64, and 78
Percent change from baseline in plasma pharmacodynamic biomarker | Days 1, 8, 29, 36, 50, 64, and 78
Absolute change from baseline in disease-specific biomarkers | Days 1, 8, 29, 36, 50, 64, and 78
Percentage change from baseline in disease-specific biomarkers | Days 1, 8, 29, 36, 50, 64, and 78
Absolute change from baseline β-Hydroxybutyrate and lipid profile | Days 1, 8, 29, 36, 50, 64, and 78
Percent change from baseline β-Hydroxybutyrate and lipid profile | Days 1, 8, 29, 36, 50, 64, and 78
Maximum observed plasma drug concentration (Cmax) | Day 1 to Day 162
Time to reach maximum observed plasma concentration (tmax) | Day 1 to Day 162
Terminal elimination rate constant, estimated by log-linear least-squares regression of the terminal part of the concentration-time curve (λz) | Day 1 to Day 162
Apparent terminal elimination half-life associated with the terminal slope (λz) of the semi-logarithmic concentration-time curve, estimated as (ln2)/λz (t½λz) | Day 1 to Day 162
Area under the plasma concentration-time curve from time zero to 48 hours after dosing (AUC(0-48h)) | Day 1 to Day 162
Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUClast) | Day 1 to Day 162
Area under the concentration-time curve from time zero extrapolated to infinity. AUC is estimated by AUClast + Clast/λz where Clast is the last observed quantifiable concentration (AUC) | Day 1 to Day 162
Apparent total body clearance of drug from plasma after extravascular administration calculated as Dose/AUC (CL/F) | Day 1 to Day 162
Mean residence time (MRT) | Day 1 to Day 162
Time delay between drug administration and the first observed concentration in plasma (tlag) | Day 1 to Day 162
Apparent volume of distribution for parent drug at terminal phase (extravascular administration), estimated by dividing the apparent clearance (CL/F) by λz (Vz/F) | Day 1 to Day 162
Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (AUClast/D) | Day 1 to Day 162
Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUC/D) | Day 1 to Day 162
Observed maximum plasma concentration divided by the dose administered (Cmax/D) | Day 1 to Day 162
Time of the last quantifiable concentration (tlast) | Day 1 to Day 162
Maximum observed plasma drug concentration at steady state (Cssmax) | Day 1 to Day 162
Minimum observed drug concentration at steady state (Cssmin) | Day 1 to Day 162
Time to reach maximum observed plasma concentration at steady state (tssmax) | Day 1 to Day 162
Area under the concentration-time curve in the dose interval (AUCss) | Day 1 to Day 162
Apparent total body clearance of drug from plasma after extravascular administration calculated as Dose/AUCss (CLss/F) | Day 1 to Day 162
Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUCss/D) | Day 1 to Day 162
Observed maximum plasma concentration divided by the dose administered (Cssmax/D) | Day 1 to Day 162
Accumulation ratio based on Cmax (RacCmax) | Day 1 to Day 162
Accumulation ratio based on AUC (RacAUC) | Day 1 to Day 162
Temporal change parameter in systemic exposure (TCP) | Day 1 to Day 162
Amount of analyte excreted into the urine from time t1 to t2 (Ae(t1-t2)) | Day 1 and Day 57: Pre-dose and between 0-6 hours, 6-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Cumulative amount of analyte excreted from time zero through the last sampling interval (Ae(0-last)) | Day 1 and Day 57: Pre-dose and between 0-6 hours, 6-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Fraction of dose excreted unchanged into the urine from time t1 to t2 (fe(t1-t2)) | Day 1 and Day 57: Pre-dose and between 0-6 hours, 6-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Cumulative fraction (%) of dose excreted unchanged into the urine from time zero to the last measured time point (fe(0-last)) | Day 1 and Day 57: Pre-dose and between 0-6 hours, 6-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Renal clearance of drug from plasma, estimated by dividing Ae(0-t) by AUC(0-t) where the 0-t interval is the same for both Ae and AUC (CLR) | Day 1 and Day 57: Pre-dose and between 0-6 hours, 6-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Change from placebo to Week 10 in PNPLA3 messenger ribonucleic acid (mRNA) and protein expression (Cohort 4 only) | Week 10
Change from baseline to Week 10 in PNPLA3 mRNA and protein expression (Cohort 4 only) | Baseline, Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, MD, MHSc, Principal Investigator — Director, NAFLD Research Center Director of Hepatology, Professor of Medicine Vice Chief, Division of Gastroenterology University of California at San Diego ACTRI Building, 1W202 9500 Gilman Drive La Jolla, CA, 92037-0887
Locations (14):
- United States (14):
  - Research Site, Chula Vista, California
  - Research Site, La Mesa, California
  - Research Site, Montclair, California
  - Research Site, San Diego, California
  - Research Site, Doral, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Morehead City, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Armisen J, Rauschecker M, Sarv J, Liljeblad M, Wernevik L, Niazi M, Knochel J, Eklund O, Sandell T, Sherwood J, Bergenholm L, Hallen S, Wang S, Kamble P, Bhat M, Maxvall I, Wang Y, Lee RG, Bhanot S, Guo S, Romeo S, Lawitz E, Fjellstrom O, Linden D, Blau JE, Loomba R. AZD2693, a PNPLA3 antisense oligonucleotide, for the treatment of MASH in 148M homozygous participants: Two randomized phase I trials. J Hepatol. 2025 Jul;83(1):31-42. doi: 10.1016/j.jhep.2024.12.046. Epub 2025 Jan 9. PMID 39798707
- [Derived] Lai M, Lai JC, Allegretti AS, Patidar KR, Cullaro G. Investigating the Association between Steatotic Liver Disease and CKD in a Nationally Representative Sample. Kidney360. 2024 Dec 1;5(12):1844-1852. doi: 10.34067/KID.0000000569. Epub 2024 Sep 5. PMID 39235870